CLINICAL TRIAL: NCT06706089
Title: Nurse-led Educational Intervention on Patients With Glaucoma With Low Health Literacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hellenic Mediterranean University (Other)
Responsible Party: Principal Investigator, Konstantinos Giakoumidakis, Associate Professor, Department of Nursing, School of Health Sciences, Hellenic Mediterranean University, Hellenic Mediterranean University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 103/08.04.2023
Record Dates: First submitted 2024-10-18; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Glaucoma; Health Literacy; Patient Activation
Keywords: Health literacy; glaucoma; patient activation; Nurse-led training intervention
MeSH Terms: conditions — Glaucoma; Patient Participation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No intervention: Control Group: Group A (N=156) (No Intervention): This group did not receive this study's intervention, and were only used for comparisons with the experimental group.
- Experimental: Group B: Intervention Group (N=156) (Experimental): This group received the described intervention of this study.
  Interventions: Other: Nurse-led educational intervention

INTERVENTIONS:
Other: Nurse-led educational intervention — This nurse-led educational intervention included: a) an oral training session regarding glaucoma by the P.I. lasting 15 minutes, b) provision of printed informational material (leaflet) and c) provision of appropriately selected free informational videos from the World Glaucoma Association on the "YouTube" -online platform. All of the above mentioned educational methods focused on the disease, its treatment and its long-term management. The oral training session took place in an appropriate, quiet and clean area, respecting the patient's privacy. During this process, study participants had the opportunity and time to ask questions and ask for clarifications or additional information.
  Arms: Experimental: Group B: Intervention Group (N=156)

SUMMARY:
Introduction: Chronic diseases are a major cause of ill health, disability and death worldwide and are potentially preventable and treatable. Glaucoma is among the main causes of morbidity and blindness; its early detection can reduce the risk of poor patient outcomes. The existence of health illiteracy among these patients and the absence of self-management of these diseases are a barrier to their effective management worldwide.

Aim: The investigation of effect of a nurse-led patient education on both the incidence of negative outcomes and the activation levels of glaucoma patients with low health literacy status. Secondary objectives of the present study are the assessment of patient activation and health literacy prior to (baseline) and after (follow-up period)patient education at predefined times, as well as the association of patient socio-demographic and clinical parameters with the patient activation and health literacy levels.

Methodology: A quasi experimental study will be conducted with follow-up in a population of patients with diagnosed glaucoma, who will attend the outpatient ophthalmological clinic of the Heraklion University General Hospital. The research tools that will be used for the assessment of health literacy will be the Greek version of the European Health Literacy Survey Questionnaire 16 (HLS-EU-16) and for the assessment of the patients' activation level the Patient Activation Measure - 13 (PAM-13) questionnaire will be used, which will be translated . The data will be analyzed using the Statistical Package for Social Sciences (SPSS) (IBM Statistics) software program, version 24.0, and ethical and moral rules will be followed.

Expected results: The proposed study is expected to underline both the level of health literacy of glaucoma patients in Greece and the importance of self-management of chronic diseases carried by patients. Additionally, the present study is expected to highlight the significance of the nurse-led education process of patients with low health literacy status on reducing the poor patient outcomes incidence and the improvement of their activation levels, leading to the optimal self-management and self-care.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Informed written consent to participate in the study
* Adequate knowledge of the Greek language (writing and reading)
* Diagnosis of the condition for at least six months

Exclusion Criteria:

* Patients with incomplete health records
* Patients who provided incomplete information
* Patients who wished to stop participating were excluded

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2023-11-20 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
Health literacy Survey Questionnaire (HLS-EU-16) | From enrollment to the end of the intervention at 6 months
  The assessment of health literacy using the Greek version of the European Health Literacy Survey Questionnaire (HLS-EU-16) is an important method for understanding participants' knowledge and skills in managing their health.
  In the HLS-EU-16, each question is scored from 1 to 4 based on how easily participants understand and apply health-related information:
  1. = Very difficult
  2. = Difficult
  3. = Easy
  4. = Very easy
  Minimum score: The lowest score is 16 (1 x 16 questions), indicating very low health literacy.
  Maximum score: The highest score is 64 (4 x 16 questions), indicating high health literacy.
  Health Literacy Levels: The total score is converted to a percentage and classified as follows:
  * Sufficient health literacy: Easily understands and applies health information.
  * Problematic health literacy: Has difficulty understanding or applying health information.
  * Inadequate health literacy: Faces major challenges using basic health information, impacting health outcomes.
Patient Activation Measure - 13 (PAM-13) | From enrollment to the end of the intervention at 6 months
  The Patient Activation Measure - 13 (PAM-13) is widely used to assess patient activation, meaning patients' willingness and ability to manage their health and make informed decisions to improve their quality of life. The PAM-13 includes 13 questions rated on a 4-point Likert scale from [1] "strongly disagree" to [4] "strongly agree," with a "not applicable" option. To calculate the PAM score, responses are summed, divided by the number of valid responses (excluding "not applicable"), and multiplied by 13. This raw score is then converted to a final score from 1 to 100 using calibration tables. Based on this score, patients are classified as follows:
  * Level 1 (≤ 47.0): Patients lack belief in activation.
  * Level 2 (47.1-55.1): Patients understand but find action difficult
    .• Level 3 (55.2-67.0): Patients actively manage their health.
  * Level 4 (≥ 67.1): Patients continue positive behaviors.

CONTACTS AND LOCATIONS:
Locations (1):
- Hellenic Mediterranean University, Heraklion, Crete, Greece